CLINICAL TRIAL: NCT07039708
Title: A Computer-based Memory Strategy Training Program to Promote Everyday Performance in Healthy Older Adults, Older Adults With Memory Complaints, Mild Cognitive Impairment and Mild Dementia
Brief Title: A Computer-based Memory Strategy Training Program for Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LIU Karen, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HongKongPU_E-MinD Life Semanti
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-06

CONDITIONS: Healthy Older Adults; Memory Complaints; Mild Cognitive Impairment (MCI)
Keywords: computer-based; memory training; activities of daily living; older adults; feasibility
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-MinD Life Semantic (Experimental): Participants receive the E-MinD Life (Semantic) programme.
  Interventions: Behavioral: E-MinD Life Semantic
- Cognitive stimulation (Active Comparator): Participants will receive cognitive stimulation.
  Interventions: Behavioral: Cognitive stimulation

INTERVENTIONS:
Behavioral: E-MinD Life Semantic — The E-MinD Life programme is designed to teach semantic memory strategies. The memory strategies are applied to 12 common daily activities required for community living, e.g. meal preparation, laundry activities, and built into the E-MinD Life programme on a computer-based platform. The intervention runs over 9 weeks with one 45-minute individual face-to-face or online healthcare-professional-led session and two 30-minute, family-assisted home sessions per week. During the home sessions, participants will complete the same activities as those learnt during the healthcare-professional-led sessions. Family members or carers will be invited to join the healthcare-professional-led sessions as observers and support the participants in the home sessions if needed.
  Arms: E-MinD Life Semantic
Behavioral: Cognitive stimulation — Participants will receive stimulation for visual attention and memory through activities such as playing a game that requires them to find missing pieces, and auditory attention and memory through activities such as remembering a song. The intervention will adopt a similar structure as the E-MinD Life Semantic group, with one 45-minute individual face-to-face or online healthcare-professional-led session and two 30-minute, family-assisted home sessions per week for 9 weeks.
  Arms: Cognitive stimulation

SUMMARY:
A computer-based cognitive rehabilitation program based on daily tasks utilising the semantic encoding strategies called Enhancing Memory in Daily Life (E-MinD Life) has been developed for Chinese people. The aim of the E-MinD Life is to delay functional deterioration associated with possible cognitive changes in healthy older adults, older adults with memory complaints, mild cognitive impairment (MCI) and mild dementia. This project will pilot-test the E-MinD Life in Chinese healthy older adults, older adults with memory complaints, MCI and mild dementia.

DETAILED DESCRIPTION:
The objectives of the study are to investigate the feasibility and pilot-test the benefits of the computer-based E-MinD Life (Semantic) program to promote everyday performance in healthy older adults, older adults with memory complaints, mild cognitive impairment (MCI) and mild dementia in Hong Kong using a randomised control trial.

Three groups of participants will be recruited: (1) 15 healthy older adults, (2) 15 older adults aged over 65 years with memory complaints, or older adults aged over 65 years, meeting the diagnostic criteria for MCI with a Clinical Dementia Rating score of 0 or having mild dementia with a Clinical Dementia Rating score of 1. All participants will have no depression and other clinical conditions that may affect their cognition. Their scores on the Montreal Cognitive Assessment will be recorded. Their carers or family members are invited to participate.

ELIGIBILITY:
Inclusion Criteria:

Group 1: healthy older adults aged 65 years or above Group 2: older adults aged 65 years or above with memory complaints Group 3: older adults aged 65 or above with mild cognitive impairment

Exclusion Criteria (for all groups 1, 2 and 3)

- have depression and other clinical conditions that may affect their cognition.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Accceptability | End of the intervention at 9 weeks
  Acceptability is measured using a structured questionnaire divided into five sections: (1) the therapist-led group sessions, (2) the self-administered individual sessions, and (3) the computer program interface and iPad usability, (4) the overall program design and structure and (5) overall satisfaction. Participants are invited to give quantitative ratings on four dimensions under each section: (a) perceived effectiveness (e.g., whether the program improved cognitive strategy use), (b) relevance (e.g., how applicable the activities were to daily life), (c) convenience (e.g., ease) and (d) clarity. Responses are collected using a 4-point Likert scale, ranging from 1 "Completely disagree" to 4 "Completely agree," with higher scores indicating greater acceptability.

SECONDARY OUTCOMES:
Feasibility by measuring the attendance rate | Through the intervention for 9 weeks, attendance at each session
  Feasibility by measuring the intervention attendance rate
Consortium to Establish a Registry for Alzheimer's Disease - Neuropsychological Assessment Battery (CERAD-NAB) | From enrollment to the end of intervention at 9 weeks
  The CERAD-NAB provides a profile on cognitive function by assessing cognitive deficits and was validated in a Chinese version. This study will use all subtests, including Verbal Fluency (J1), Boston's Naming (J2), Mini-Mental State Examination (MMSE, J3), Word List Memory (J4), Constructional Praxis (J5), Word List Recall (J6), Word List Recognition (J7) and Recall of Constructional Praxis (J8). The total score ranges from 0 -115 with a higher score indicating better performance.
Digit Span Test | From enrollment to the end of intervention at 9 weeks
  The Digit Span Test consists of Digit Span Forward (DSF) and Digit Span Backward (DSB), measures immediate verbal recall, attentional capacity and working memory. The score is the number of digits in the longest successfully recalled sequence. A higher score indicates a better performance.
Lawton Instrumental Activities of Daily Living Scale | From enrollment to the end of intervention at 9 weeks
  The self-reported Lawton Instrumental Activities of Daily Living Scale-Chinese version (IADLS) assesses one's ability to independently perform eight domains of instrumental daily activities such as meal preparation, laundry work, and shopping. The scale consists of nine items, each rated on a 3-point or 4-point scale, with a total score ranging from 0 to 18 or higher. A higher score indicates a better performance
Disability Assessment for Dementia (DAD) | From enrollment to the end of intervention at 9 weeks
  The Chinese version of the Disability Assessment for Dementia (DAD) is a survey, completed by a proxy/carer, that evaluates the level of independence in daily activities for a person who has dementia or cognitive impairment. The DAD is scored based on a "yes/no" system, where "yes" indicates the person performed the activity without help, and "no" indicates they did not. The number of "yes" responses is totalled, and then converted to a percentage score out of 100. Higher percentage scores indicate better functional ability.
EuroQoL- 5 Dimensions - 5 Levels Hong Kong version (EQ-5D-5L_HK) | From enrollment to the end of intervention at 9 weeks
  The EQ-5D-5L HK measures health-related quality of life in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, using five rating levels (33). The 5-level health status is converted to a utility value, ranging from 0 (death) to 1 (full health). The EQ-5D-5L HK includes a Visual Analogue Scale where respondents rate their overall health on a scale of 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Liu, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The project is applying for external funding. The IPD will not be shared at this stage.